CLINICAL TRIAL: NCT02863627
Title: What Care Pathways for Newborns Consulting Pediatric Emergencies? Prospective Study Over One Year Newborn Pediatric Emergencies (NNUP)
Brief Title: What Care Pathways for Newborns Consulting Pediatric Emergencies? Prospective Study Over One Year
Acronym: NNUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-HPNCL-04
Record Dates: First submitted 2016-06-28; First posted 2016-08-11 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Emergencies
Keywords: Emergencies; newborn; care
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Newborn Care Pathway (Experimental): two telephone interviews conducted after the emergency department visit will be used to gather data to meet the objectives of this study.
  Interventions: Other: Newborn Care Pathway

INTERVENTIONS:
Other: Newborn Care Pathway — consultation with the pediatric emergency, two telephone interviews to complete Questionnaires with the parents after the emergency department visit

SUMMARY:
This study will evaluate the course of care of newborns, to understand why some newborns have improper care pathways, particularly as regards the first medical consultation at the exit of motherhood. It is also to organize a better quality care network to hospital discharge to avoid unnecessary use of pediatric emergencies, which represents a real public health problem.

DETAILED DESCRIPTION:
In 2014, newborns represented 1.57% of passages (or 906 newborns) of Emergency Pediatric Hospitals CHU de Nice-Lenval. This proportion is significant and steadily increasing (2013: 820 newborns or 1.46% of passes). The experienced team of pediatric emergency is that the majority of consultations respite care and child care could well be managed city. The bibliographic data confirms this feeling.

But no study has examined the course of care of the newborn during its first month of life. In 2014, in its recommendations for good practice for the release of motherhood after giving birth, the HAS recommends a medical examination by a pediatrician (or a general practitioner with experience of pathologies of the newborn) between 6 and 10 days of life. Other consultations (midwife, health visitor in PMI) is not required. Moreover, in its brochure to mothers, prompt medical attention is recommended in certain situations (fever, vomiting ...) but without specifying the organization. The pediatric emergency therefore no place, except for emergencies, in the course of care of newborns. But the care pathway proposed by the HAS is it feasible? And it reduces unnecessary use of pediatric emergency?

The main objective of this study is to evaluate the course of care of newborns consultant pediatric emergency looks to the recommendations of the 2014 HAS.

The secondary objectives are:

* Identify factors associated with abnormal care course and / or consultation with appropriate non emergencies.
* Evaluate the reasons why parents of newborns to consult pediatric emergency first-line concern and before / after the emergency department visit.
* Evaluate the information received by parents on maternity or during medical consultations or previous paramedical.

The primary endpoint is the assessment of the course of care of newborns consultant pediatric emergencies of appropriately (that is to say addressed newborn and / or implementation of additional tests and / or hospitalization) or not adapted.

The secondary endpoints are:

* Description of clinical and demographic characteristics of the newborn, the social characteristics of the parents.
* Description of the consultation to pediatric emergencies.
* Information Evaluation received by parents on the time of the first medical consultation at the exit of motherhood and the reason for consultation to pediatric emergencies.

This is a biomedical intervention study Routine care, single-center prospective, non-randomized. Will be included all newborns (that is to say, child ≤ 28 days of life) consultant to hospital emergency NICE-Lenval Hospital, and after obtaining the non-opposition of the two parents. The number of patients needed is 280 newborns. The duration of inclusion is one year.

Following consultation with the pediatric emergency, parents will be contacted 2 times:

* 2-7 days after the consultation: clinical and demographic characteristics of the newborn, social characteristics of parents, information received by parents, whether (s) consultation (s) Medical (s) or paramedic (s) already completed and anxiety parents before / after the emergency department visit.
* In the week following the first month of life the child complete the child care course.

The data on emergency department visit (which made additional tests and fate of the child) will be collected from the host software pediatric emergencies.

This study will evaluate the course of care of newborns, to understand why some newborns have improper care pathways, particularly as regards the first medical consultation at the exit of motherhood.

ELIGIBILITY:
Inclusion Criteria:

* Newborn within 28 days included
* Subjects affiliated to Social Security.
* Non-opposition form signed by the two parents.

Exclusion Criteria:

* Parental refusal
* non opposition form not signed by the parents.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01-31 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation course of care of newborns | baseline
  Evaluate the course of care of newborns consultant pediatric emergencies as recommended by the National Health Authority in 2014.

SECONDARY OUTCOMES:
Evaluation of abnormal care path | baseline
  description of factors associated with abnormal care path not adapted to emergencies.
Evaluate reasons to come to pediatric emergency | baseline
  Evaluate the reasons why parents of newborns consult pediatric emergency in first intention
Evaluate the information received by parents | baseline
  Evaluate the information received by parents on maternity or during medical consultations or previous paramedical

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure HERISSE, MD, Principal Investigator — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-LENVAL, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran A, Herisse AL, Isoardo M, Valo P, Maillotte AM, Haas H, Donzeau D, Freyssinet E, Pradier C, Gentile S. Evaluation of compliance with early postbirth follow-up and unnecessary visits to the paediatric emergency department: a prospective observational study at the Lenval Children's Hospital in Nice. BMJ Open. 2022 Jan 6;12(1):e056476. doi: 10.1136/bmjopen-2021-056476. PMID 34992122